CLINICAL TRIAL: NCT04221061
Title: A Pilot Study Evaluating in Vivo PARP-1 Expression with18F-FluorThanatrace Positron Emission Tomography (PET/CT) in Glioblastoma
Brief Title: 18F-FluorThanatrace (PET/CT) in Glioblastoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Companion treatment trial closed early with negative results. No imaging study participants completed the full study imaging planned due to logistical difficulties.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 833963
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-surgical candidates (Other): In this arm, subjects that do not have a clinical indication for surgical resection of the recurrent tumor will start TTFields therapy 5-7 days prior to starting oral niraparib (a PARP inhibitor).
  Interventions: Drug: 18F-FluorThanatrace
- Surgical candidates (Other): In this arm, subjects who have a clinical indication for surgical resection of the recurrent tumor will receive TTFields therapy for 5-7 days prior to planned surgical resection, undergo resection, and then resume TTFields therapy and initiate niraparib post-operatively.
  Interventions: Drug: 18F-FluorThanatrace

INTERVENTIONS:
Drug: 18F-FluorThanatrace — 18F-FluorThanatrace is a novel radiopharmaceutical which measure PARP-1 expression using a Positron Emission Tomography (PET/CT) scan.
  Other Names: FTT

SUMMARY:
The subject will be a candidate for this imaging study because they have agreed to participate in a treatment study involving TTFields (Optune device), a device that uses low intensity, wave like electrical fields, and a PARP inhibitor drug (niraparib). The research study is being conducted to test how a new radioactive imaging drug called 18F-Fluorthanatrace (18F-FTT) can be used to image sites of recurrent brain cancer before or after new treatment or surgery. 18F-FTT is a drug used with an imaging test called Positron Emission Tomography/Computed Tomography (PET/CT).

DETAILED DESCRIPTION:
Participants will undergo up to three [18F]FTT PET/CT scans at the following time points:

* Baseline: Subjects from either cohort may agree to undergo a baseline [18F]FTT PET/CT prior to the start of TTFields therapy to measure baseline FTT uptake. This scan is not required and may be omitted at the discretion of the investigator or based on subject availability.
* Post-TTFields: Subjects from both cohorts will undergo an [18F]FTT PET/CT scan 3-7 days after initiation of TTFields therapy and before surgical resection or initiation of niraparib. This scan will measure the FTT uptake after TTFields therapy is initiated. This scan is required.
* Post-PARPi: Subjects from Cohort A may agree to undergo an post-therapy [18F]FTT PET/CT scan 1- 21 days after the initiation of niraparib to collect pilot data on the changes in FTT uptake after TTFields and niraparib combination therapy. This scan is not required and may be omitted at the discretion of the investigator or based on subject availability.

For each [18F]FTT PET/CT imaging session, participants will undergo approximately 60 minutes of dynamic brain scanning starting nearly simultaneously with the injection of [18F]FTT. A second optional brain scan will be done at approximately 90 minutes post-injection. Each imaging session will include an injection of up to 12 mCi (approximate range for most studies is anticipated to be 8-12 mCi) of [18F]FTT.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 22 years of age
2. Participants will have a diagnosis of glioblastoma and be enrolled in the companion treatment trial, IRB 832694.
3. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of childbearing potential at screening.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.

Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Evaluate uptake of [18F]FTT in recurrent glioblastoma after initiation of TTFields therapy. | 3 years
  Evaluate uptake of [18F]FTT in recurrent glioblastoma after initiation of TTFields therapy.

SECONDARY OUTCOMES:
Correlate [18F]FTT uptake measures with Homologous recombination deficiency (HRD) status or other markers of "BRCAness". | 3 years
  Correlate [18F]FTT uptake measures with Homologous recombination deficiency (HRD) status or other markers of "BRCAness".
  To determine pre-/post-treatment changes in [18F]FTT uptake after initiation of TTFields therapy.
  To determine pre-/post-treatment changes in [18F]FTT uptake after initiation of PARP inhibitor.
  To correlate PARP expression by pathology testing with uptake of [18F]FTT in surgical subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Austin R Pantel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States